CLINICAL TRIAL: NCT03493594
Title: Effectiveness of a Community Based Early Nutrition Program on Promoting Breastfeeding and Optimizing Infant Growth and Diet Quality
Brief Title: Effectiveness of an Early Nutrition Program on Promoting Breastfeeding and Optimizing Infant Growth and Diet Quality
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Man-sau WONG, Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CUHKFSTRC2018-01
Record Dates: First submitted 2018-03-20; First posted 2018-04-10 (Actual); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Breastfeeding; Infant Development
Keywords: Early nutrition; Breastfeeding; Infant growth
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Control group will receive standard health care.
  To improve the compliance of the subjects, both intervention group and control group can attend one vision development workshop at 2-month postpartum and two parenting workshops at 6- and 12-month postpartum.
- Nutrition education program (Experimental): The intervention group will receive an early nutrition program for 12 months. Workshops format will be mainly in form of talks and experience sharing groups which run by lactation consultants, nutritionists / dietitians. All classes and workshops will be run for 4-6 times to cater for subjects recruited in different phases.
  To improve the compliance of the subjects, both intervention group and control group can attend one vision development workshop at 2-month postpartum and two parenting workshops at 6- and 12-month postpartum.
  Interventions: Other: Nutrition education program

INTERVENTIONS:
Other: Nutrition education program — online platform support, workshop, seminar and cooking demo etc
  Arms: Nutrition education program

SUMMARY:
Effective early life programs that reduce the long-term non-communicable diseases (NCDs) risk could bring great economic benefits to the society. However, there is a lack of local data on the effect of nutrition on child growth and most research on early life intervention focus on disease models such as obese women to improve offspring health outcomes. There is limited research on postpartum interventions in the community that optimize maternal and infant nutrition through improving success of breastfeeding, infant growth diet quality and microbiota to enhance health in the adulthood.

In this study, it is hypothesized that our early nutrition program could promote breastfeeding successful rate (increase the number of months the mothers breastfed their infants) and improve growth status, diet quality and microbiota of the infants which may reduce the risk of NCDs in the adulthood. The planned project proposal would like to include 240 pairs of mothers and infants. In order to test the protocol in the planned proposal, the investigators hope to run a pilot study to set up this community based early nutrition program including breastfeeding workshops and supports, healthy lifestyle courses, parenting education, introduction of solid foods for infants, child development and cooking classes of infant foods. the investigators will evaluate the effectiveness of this early nutrition program and determine its impacts on breastfeeding, infant growth (by comparing infants' biomarkers and microbiota in different stages) , diet quality and microbiota, as well as the benefits to the postpartum mothers such as reducing the postpartum weight retention so that to generate pilot result and facilitate the up scale study that the investigators proposed in the planned proposal.

The ultimate goal is that a long term follow up with the children in this project could also be arranged to determine the long term health effects of this early nutrition program.

DETAILED DESCRIPTION:
Study background:

Effective early life programs that reduce the long-term non-communicable diseases (NCDs) risk could bring great economic benefits to the society. NCDs are responsible for roughly two-thirds of worldwide death and cause large burden of health care cost. Most policies nowadays that combat disease focus on treatment after disease occurs and on reducing risk factors in adult life. Early life interventions are an unexplored and promising new avenue of health policy . One of the oldest US early life intervention programs, the Carolina Abecedarian Project, started from 1970s has been shown to have substantial benefits in boosting adult health. However, most research on early life intervention focus on disease models such as obese women to improve offspring health outcomes. There is limited research on postpartum interventions in the community that optimize maternal and infant nutrition through improving success of breastfeeding, infant growth, diet quality and microbiota to enhance health in the adulthood

Aim of study:

To evaluate the effects of postpartum nutrition program on i) success of breastfeeding by comparing the average duration of breastfeeding between intervention group and control group (primary outcome) ii) diet quality of the infants and mothers (secondary outcome) The diet quality will be measured by 3-day dietary records using Diet Quality Index-International (DQI-I).

Briefly, the DQI-I assesses four categories (variety, adequacy, moderation, and overall balance) and contains six food items and 11 nutrient items. This scoring scale is complex. The maximum possible score for each category ranges from 10 to 40 points, and the full score is 100 points.

Paired t-tests will be used to compare the difference between intervention group and control group.

iii) the infant growth by comparing the Z-scores of weight-for-age, length-for-age, BMI-for-age and head circumference-for-age at 2, 4, 6, 8, 10 and 12 month old between intervention group and control group (secondary outcome) Z-score (or SD-score) = (observed value - median value of the reference population) / standard deviation value of reference population

iv) the microbiota profiles (secondary outcome)

Method of Investigation:

In this project, a randomized controlled trial will be conducted which subjects will be 40 pairs of local Chinese healthy postpartum mothers aged 18-40 years old and their infants. The participants will be randomly assigned into 1:1 ratio to the control group or the intervention group. A study coordinator will randomize subjects by means of a computer-generated list of random numbers in blocks of 4. Treatment assignments will be concealed in consecutively-numbered sealed envelopes, which will be opened sequentially upon subject enrollment.

ELIGIBILITY:
Inclusion Criteria for mothers:

* Postpartum mothers: Aged 18-40 years old
* Hong Kong residents having resided in Hong Kong for a continuous period of not less than 18 months
* vaginal delivery at full term (>37 gestation weeks)
* first pregnancy and give birth to singleton infant

Inclusion Criteria for Infants:

* Full term
* Born by vaginal delivery (>37 gestation weeks)
* singleton infant with no known abnormality.

Exclusion Criteria:

* Concurrent participation in any clinical trial or study
* Complicated pregnancy such as preeclampsia and gestational diabetes
* Special dietary restrictions for examples gluten-free diets, vegan or any restrictions due to food allergies;
* Suffer from renal, liver or thyroid dysfunction, cognitive impairment, or any other indication of a major medical or psychological illness, as judged by the investigators as ineligible to participate the study.

Max Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — the subjects are mothers and their infants so Female subjects needed to be selected while there is no sex limitation in the infants
Enrollment: 96 (Estimated)
Dates: Start 2018-04-16 (Estimated); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
Success rate of breastfeeding | through study completion, an average of 1 year
  success rate of breastfeeding by comparing the average duration of breastfeeding

SECONDARY OUTCOMES:
Diet quality | through study completion, an average of 1 year
  Diet quality of the infants and mothers at 2, 4, 6, 8, 10 and 12 month old
Infant growth | through study completion, an average of 1 year
  Infant growth by comparing the Z-scores of weight-for-age, length-for-age, BMI-for-age and head circumference-for-age at 2, 4, 6, 8, 10 and 12 month old
Microbiota profiles | through study completion, an average of 1 year
  Microbiota profiles at 2, 4, 6, 8, 10 and 12 month old

CONTACTS AND LOCATIONS:
Overall Officials: Man-sau Wong, PhD, Principal Investigator — The Hong Kong Polytechnic University

IPD SHARING:
Plan to Share IPD: No